CLINICAL TRIAL: NCT03015727
Title: Induction Chemotherapy With Docetaxel and Cisplatin Followed by Radiotherapy Alone or Concurrent Chemoradiotherapy in Locally Advanced Nasopharyngeal Carcinoma
Brief Title: Induction Chemotherapy Followed by Radiotherapy Alone or Concurrent Chemoradiotherapy in Nasopharyngeal Carcinoma
Acronym: IRCNPC
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Zhejiang Cancer Hospital (Other)
Collaborators: Zhejiang Provincial People's Hospital (Other); The Central Hospital of Lishui City (Other); Jinhua Central Hospital (Other); First Affiliated Hospital of Wenzhou Medical University (Other); Ningbo Medical Center Lihuili Eastern Hospital (Unknown); People's Hospital of Quzhou (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ZhejiangCH 01536224
Record Dates: First submitted 2016-12-24; First posted 2017-01-10 (Estimated); Last update posted 2017-01-10 (Estimated); Status verified 2016-12

CONDITIONS: Locally Advanced Nasopharyngeal Carcinoma
Keywords: nasopharyngeal carcinoma; Induction chemotherapy; radiotherapy; chemoradiotherapy
MeSH Terms: conditions — Nasopharyngeal Carcinoma | interventions — Docetaxel; Cisplatin; Drug Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- IC+RT group (Experimental): 3 cycles of TP neoadjuvant chemotherapy at day1,22 and 43 with docetaxel 75mg/m2 and cisplatin 75mg/m2. And then radiation using IMRT/TOMO without concurrent chemotherapy.
  Interventions: Drug: Docetaxel; Drug: Cisplatin; Radiation: IMRT/TOMO
- IC+CCRT group (Active Comparator): 3 cycles of TP neoadjuvant chemotherapy at day1,22 and 43 with docetaxel 75mg/m2 and cisplatin 75mg/m2.And then chemoradiation using IMRT/TOMO with 2 cycles of cisplatin concurrent chemotherapy at 100mg/m2.
  Interventions: Drug: Docetaxel; Drug: Cisplatin; Radiation: IMRT/TOMO; Drug: Chemotherapy

INTERVENTIONS:
Drug: Docetaxel — 3 cycles of DOC neoadjuvant chemotherapy at day1,22 and 43 with docetaxel 75mg/m2.
  Other Names: DOC
Drug: Cisplatin — 3 cycles of DDP neoadjuvant chemotherapy at day1,22 and 43 with cisplatin 75mg/m2.
  Other Names: DDP
Radiation: IMRT/TOMO — intensity modulated radiation therapy or tomotherapy
Drug: Chemotherapy — 2 cycles of cisplatin concurrent chemotherapy at day 64 and 85 with cisplatin 100mg/m2.
  Other Names: concurrent chemotherapy
  Arms: IC+CCRT group

SUMMARY:
In this study, the investigators aim to compare the progression-free survival (PFS) and side effects of radiotherapy (RT) and concurrent chemoradiotherapy (CCRT) in locoregionally advanced nasopharyngeal carcinoma (NPC) patients with a satisfactory tumor response (complete response or partial response) after neoadjuvant chemotherapy (NACT).

DETAILED DESCRIPTION:
In this study, the investigators aim to compare the survival outcomes and side effects of radiotherapy (RT) and concurrent chemoradiotherapy (CCRT) in locoregionally advanced nasopharyngeal carcinoma (NPC) patients with a satisfactory tumor response (complete response or partial response) after neoadjuvant chemotherapy (NACT) with Docetaxel and Cisplatin treated using intensity-modulated radiotherapy (IMRT) or tomotherapy (TOMO).

ELIGIBILITY:
Inclusion Criteria:

1. Patients with newly histologically confirmed non-keratinizing carcinoma.
2. Tumor staged as N2-3 or T3-4 (according to the 7th AJCC staging system)
3. No evidence of distant metastasis (M0)
4. Performance status: KPS>70
5. With normal liver function test (ALT, AST <1.5ULN)
6. Renal: creatinine clearance >60ml/min
7. Without hematopathy,marrow: WBC >4*109/L, HGB>80G/L, and PLT>100*109/L.
8. With controlled blood glucose for diabetes patients
9. Written informed consent
10. satisfactory tumor response (complete response or partial response) after neoadjuvant chemotherapy (NACT)

Exclusion Criteria:

1. WHO type I squamous cell carcinoma or adenocarcinoma
2. Age >65 or <18
3. With a history of renal disease
4. Prior malignancy (except adequately treated carcinoma in-situ of the cervix or basal/squamous cell carcinoma of the skin)
5. Previous chemotherapy or radiotherapy (except non-melanomatous skin cancers outside the intended RT treatment volume)
6. Patient is pregnant or lactating
7. Peripheral neuropathy
8. Emotional disturbance

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 440 (Estimated)
Dates: Start 2016-12; Primary Completion 2022-12 (Estimated); Study Completion 2024-12 (Estimated)

PRIMARY OUTCOMES:
Progress Free Survival (PFS) | 3 years after the inception assignment
  PFS means assignment to the date of any local or distant progress of the disease.

SECONDARY OUTCOMES:
Overall Survival (OS) | 3 years and 5 years after the inception of the assignment
  The overall survival denote to assignment to date of death from any cause.
Adverse Events | Participants will be followed for the duration of hospital stay, an expected average of 100 days and every 3 months thereafter for 5 years
  Observe and record the toxicity profile (including but not limit to mucositis, liver and kidney function, et al.) according NCI-CTCAE (3rd edition) during the neoadjuvant chemotherapy, chemoradiation and follow-up.

CONTACTS AND LOCATIONS:
Overall Officials: Xiaozhong Chen, Study Chair — Zhejiang Cancer Hospital
Locations (1):
- Xiaozhong Chen, Hangzhou, Zhejiang, China

IPD SHARING:
Plan to Share IPD: Undecided